CLINICAL TRIAL: NCT00799071
Title: Investigation of POsaconazole Prophylaxis in Children With Chronic Granulomatous Disease (CGD): Pharmacokinetics and Tolerability (iPOD)
Brief Title: Pharmacokinetics of Posaconazole in Children With Chronic Granulomatous Disease (CGD)
Acronym: iPOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCN-AKF 08.01
Record Dates: First submitted 2008-11-26; First posted 2008-11-27 (Estimated); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Chronic Granulomatous Disease
Keywords: prophylaxis; CGD; pharmacokinetics
MeSH Terms: conditions — Granulomatous Disease, Chronic | interventions — posaconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- posaconazole (Experimental): posaconazole as antifungal prophylaxis
  Interventions: Drug: posaconazole (PSZ)

INTERVENTIONS:
Drug: posaconazole (PSZ) — Intake of PSZ oral suspension 40mg/ml twice daily with food. Starting dose is based on bodyweight. The dosage will be adjusted if the exposure is not adequate based on PSZ trough level on Day 10 and 20.
  Other Names: Noxafil

SUMMARY:
The purpose of this study is to find a dose for a twice daily regimen for posaconazole (PSZ) as prophylactic treatment in children with CGD, based on the PSZ trough level.

DETAILED DESCRIPTION:
At this moment itraconazole is the drug of first choice in the prophylaxis of fungal infections in children with CGD. Breakthrough fungal infections while on itra-conazole prophylaxis are described in literature indicating the need for a drug with a broader antifungal spectrum. PSZ might provide in this need. PSZ may also have a clinical safety and tolerability advantage over other antifungal agents. Because PSZ is metabolized through phase II glucuronidation it is less common to be subject to drug interactions. PSZ is known to be a CYP3A4 inhibitor, but does not inhibit other CYP enzymes, therefore it may exhibit fewer drug interactions as compared with other azole antifungal agents.

Treatment of children is still off-label use. No data have been published to date on the exposure of PSZ in children under the age of 8 or in children with CGD. There is an urgent need to study the use of PSZ in these young children. Furthermore, the current regimen for antifungal prophylaxis requires a three times daily administration of PSZ. For this specific purpose less complex dosing schedules are warranted thus defining the need to examine a twice daily schedule.

As the tolerability and pharmacokinetics are unknown in patients under the age of 8 years and only limited data are available for age groups 8 to 16 years, we propose a feasibility study of a twice daily regimen of PSZ prophylaxis in CGD patients. With this information available we can suggest a dosage for future prophylaxis in this patient group.

ELIGIBILITY:
Inclusion Criteria:

* Patient has CGD, rendering him/her at risk for invasive fungal infections hence requiring antifungal prophylaxis.
* Patient is at least 2 years of age and younger than 17 years of age on the day of the first dosing.
* Parents or legal representative, and children where appropriate, willing and able to give informed consent.

Exclusion Criteria:

* Patient is suspected of an invasive fungal infection.
* Therapy with any medicinal product for which an effect on PSZ is expected. If patient is undergoing therapy with any medicinal product which may be effected by PSZ, the patient is included on condition that the investigator judges that the effects are not clinically relevant. This should be clearly recorded.
* Documented history of sensitivity/idiosyncrasy to PSZ.
* Results of serum biochemistry and hematology testing are not higher than 3x the upper limit of normal. If the results exceed these limits, the patient is included on condition that the investigator judges that the deviations are not clinically relevant. This should be clearly recorded.
* Relevant history or current condition that might interfere with drug absorption, distribution, metabolism or excretion.
* Relevant history or presence of cardiovascular disorder or renal and hepatic disorder.
* History of or current abuse of drugs, alcohol or recreational substances.
* Participation in a trial with an investigational drug within 60 days prior to the first dose.

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Posaconazole trough levels | Day 10; 20; 30

SECONDARY OUTCOMES:
adverse events monitoring | entire study

CONTACTS AND LOCATIONS:
Overall Officials: David M Burger, PharmD PhD, Principal Investigator — Radboud University Medical Centre Nijmegen
Locations (2):
- Netherlands (2):
  - Radboud University Medical Centre Nijmegen, Nijmegen, Gelderland
  - AMC, Amsterdam

REFERENCES:
- [Result] Welzen ME, Bruggemann RJ, Van Den Berg JM, Voogt HW, Gilissen JH, Pajkrt D, Klein N, Burger DM, Warris A. A twice daily posaconazole dosing algorithm for children with chronic granulomatous disease. Pediatr Infect Dis J. 2011 Sep;30(9):794-7. doi: 10.1097/INF.0b013e3182195808. PMID 21772229
- See also: Pediatr Infect Dis J. 2011 Sep;30(9):794-7. A twice daily posaconazole dosing algorithm for children with chronic granulomatous disease. — http://journals.lww.com/pidj/Abstract/2011/09000/A_Twice_Daily_Posaconazole_Dosing_Algorithm_for.18.aspx